CLINICAL TRIAL: NCT00738777
Title: A Randomized, Prospective Trial of 2-6 Weeks Pre-operative Hormonal Treatment for Hormone Receptor Positive Breast Cancer: Anastrozole +/- Fulvestrant or Tamoxifen Exposure - Response in Molecular Profile (AFTER-study).
Brief Title: Pre-operative Hormonal Treatment for Hormone Receptor Positive Breast Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: in preparation for an amendment
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: N08AFT; EudraCT; 2008-000644-13
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: pre-operative; endocrine treatment; drug resistance
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Anastrozole
  Interventions: Drug: Anastrozole
- 2 (Experimental): Anastrozole + Fulvestrant
  Interventions: Drug: Anastrozole+Fulvestrant
- 3 (Active Comparator): Tamoxifen
  Interventions: Drug: Tamoxifen
- 4 (Other): Tamoxifen (pre-menopausal and male patients)
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — 1 mg,QD,PO
  Arms: 1
Drug: Anastrozole+Fulvestrant — Anastrozole; 1 mg, QD, PO Fulvestrant; 500 mg, IM, day 1, 15, 29 and monthly thereafter
  Arms: 2
Drug: Tamoxifen — loading dose of 40 mg, TID, PO, during 7 days, Thereafter 20 mg, QD, PO
  Arms: 3
Drug: Tamoxifen — loading dose of 40 mg, TID, PO, during 7 days, Thereafter 20 mg, QD, PO
  Arms: 4

SUMMARY:
To investigate prospectively whether short term endocrine treatment can induce molecular changes, predictive for therapy response.

DETAILED DESCRIPTION:
We will perform a randomized, open-label, single-institution study. It will compare the efficacy of three different endocrine treatment regimens (Anastrozole +/- Fulvestrant or Tamoxifen) in changing proliferation-index and inducing apoptosis during a 2-6 week pre-operative treatment period in breast cancer patients. These results will be correlated to gene expression profiles, phosphorylation status of the ER, SNPs in CYP450 sequences, tamoxifen metabolite concentrations, changes in estrogen serum levels and protein expression patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven invasive adenocarcinoma of the breast
* Any tumor with a size ≥ 1cm (NOT inflammatory breast cancer)
* WHO-performance score 0 or 1
* Written informed consent

Exclusion Criteria:

* Clues of metastatic disease by clinical examination according to most recent NABON guidelines
* Multicentric breast cancer
* Inflammatory breast cancer
* Hormone replacement during the last 12 months
* Other systemic treatment during the waiting time till surgery
* Already planned date for surgery within the next 2 weeks
* Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol
* Patient's refusal to undergo a core biopsy procedure of the primary tumor before the start of treatment

NB: a concomitant malignancy within the last five years is not an exclusion criterium, because survival is not the primary endpoint. Just as prior invasive breast cancer or DCIS within the last 15 years is not an exclusion criterium.

NB: Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-07 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Decrease in tumor cell proliferation and induced apoptosis. | At baseline and after 2-6 weeks of endocrine treatment

SECONDARY OUTCOMES:
Comparison of changes in gene expression after different endocrine treatment exposures | At baseline and after endocrine treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabine C Linn, MD, Principal Investigator — NKI-AvL
Locations (4):
- Netherlands (4):
  - Medisch Centrum Haaglanden, The Hague, South Holland
  - NKI-AVL, Amsterdam
  - St. Antonius ziekenhuis, Nieuwegein
  - UMC St. Radboud, Nijmegen

REFERENCES:
- [Derived] Reinema FV, Sweep FCGJ, Adema GJ, Peeters WJM, Martens JWM, Bussink J, Span PN. Tamoxifen induces radioresistance through NRF2-mediated metabolic reprogramming in breast cancer. Cancer Metab. 2023 Feb 8;11(1):3. doi: 10.1186/s40170-023-00304-4. PMID 36755288